CLINICAL TRIAL: NCT05153772
Title: A Phase 2 Open Label Study to Evaluate the Safety and Effectiveness of 212Pb-DOTAMTATE in Subjects With Somatostatin Receptor Expressing Neuroendocrine Tumors
Brief Title: Targeted Alpha-emitter Therapy of PRRT Naïve and Previous PRRT Neuroendocrine Tumor Patients
Acronym: ALPHAMEDIX02
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Orano Med LLC (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Alphamedix-02
Record Dates: First submitted 2021-11-04; First posted 2021-12-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Neuroendocrine Tumors
Keywords: Pb212-DOTAMTATE; alpha-emitter-therapy; neuroendocrine tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pb212-DOTAMTATE (Experimental): investigational radiotherapeutic drug targeting somatostatin receptor-positive neuroendocrine tumors in PRRT naive patients (Cohort 1) and previous PRRT patients (Cohort 2)
  Interventions: Drug: AlphaMedix

INTERVENTIONS:
Drug: AlphaMedix — 212Pb-DOTAMTATE is a radiolabeled derivative of octreotide targeting somatostatin positive neuroendocrine tumors
  Other Names: Pb212-octreotide analog

SUMMARY:
Multicenter Phase 2 study of 212Pb-DOTAMTATE enrolling adult subjects with positive somatostatin positive neuroendocrine tumors with either no prior history of peptide receptor radionuclide therapy (PRRT naive) or prior history of peptide receptor radionuclide therapy (Previous PRRT)

DETAILED DESCRIPTION:
In this open-label, multicenter, single-arm Phase 2 study, adult subjects with histologically confirmed NETs and positive somatostatin analog imaging, with either no prior PRRT (PRRT naive) or prior history of peptide receptor radionuclide therapy (previous PRRT) will be enrolled to receive 212Pb-DOTAMTATE 67.6 μCi/kg dose per cycle

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years old with unresectable or metastatic histologically confirmed NET
* Subjects must have received and progressed following somatostatin analog administration
* For PRRT naive subjects, documented progression of disease following previous therapy within 12 months prior to enrollment and the presence of at least 1 site of measurable disease per RECIST 1.1
* Subjects who previously received PRRT must have documented progression of disease and at least 1 site of measurable disease per RECIST 1.1 after receiving up to 4 doses (≤ 880 mCi) of 177Lu-DOTATATE/DOTATOC and received their last dose at least 6 months prior to Day 1
* Confirmed presence of somatostatin receptors on all lesions including the non-target and measurable lesions documented by CT/MRI scans, based on positive 68Ga-DOTATATE (NETSPOT®), 64Cu-DOTATATE (Detectnet™), or other Food and Drug Administration (FDA) approved SSTR PET/CT imaging within 6 weeks prior to enrollment. Follow up imaging should be performed with the same agent or modality used at baseline;

  1. Target lesions must be positive (greater than grade 2 uptake Krenning Score) or must have a standardized uptake value of more than the normal liver background.
  2. Lytic bone lesions, with an identifiable soft tissue component, evaluated by CT or MRI, can also be considered measurable lesions if the soft tissue component otherwise meets the definition of measurability according to RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) status 0-2;
* Life expectancy of at least 12 weeks in the opinion of the investigator at the time of screening;
* Sufficient bone marrow capacity and organ function in the recent blood tests within 3 weeks prior to Day 1, as defined by:

  1. White blood cell (WBC) ≥2,500/ mm3;
  2. Absolute neutrophil count (ANC) ≥1000/mm3;
  3. Platelets ≥100,000/mm3;
  4. Hemoglobin (HgB) ≥9.0 g/dL;
  5. Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤3 X upper limit of normal (ULN);
  6. Total Bilirubin: ≤2 X ULN;
  7. Serum creatinine ≤1.7 mg/dL for PRRT naïve subjects; ≤ ULN for previous PRRT subjects;
  8. Serum albumin ≥3.0 g/L; if lower than 3.0 g/L requires normal range prothrombin time (PT) and international normalized ratio (INR), and
* Be willing to practice the following medically acceptable methods of birth control (both women of childbearing potential (WOCBP) and men who have partners of childbearing potential) from the Screening Visit through 3 months after the final administration 212Pb-DOTAMTATE

Exclusion Criteria:

* Prior whole-body radiotherapy or PRRT using 177Lu/90Y/111In-DOTATATE/ DOTATOC or Targeted Alpha Therapy (TAT).
* For subjects who previously received PRRT, prior treatment with: Prior treatment with 90Y- DOTATATE/ DOTATOC, 225Ac-DOTATATE/DOTATOC, and/or 111In-DOTATATE/ DOTATOC
* Prior regional hepatic radionuclide therapy within 4 months prior to enrollment or prior nonradioactive regional hepatic therapy within 6 months prior to enrollment.
* Known hypersensitivity to somatostatin analogues, Amino Acid infusion, or 212Pb-DOTAMTATE;
* Therapeutic use of any somatostatin analogue, including Sandostatin® LAR (within 28 days) and Sandostatin® (within 1 day) prior to Cycle 1 Day 1;
* History of myelodysplastic syndrome (MDS);
* Female subjects who are pregnant or lactating;
* Indication for surgical lesion removal with curative potential;
* Known brain metastases, unless these metastases have been treated and/or stable for 6 months prior to enrollment;
* Experimental cancer treatments or other investigational therapies within 6 weeks or five half-lives of the investigational medication prior to Day 1;
* Uncontrolled congestive heart failure (NYHA II, III, IV);
* Uncontrolled diabetes mellitus as defined by a hemoglobin A1C >10.0;
* Evidence of renal obstruction based on Tc-99m DTPA or TER for MAG3 renal scintigraphy or renal ultrasound.
* Known or active human immunodeficiency virus (HIV) or hepatitis B or C virus unless cured;
* Known or suspected active drug or alcohol abuse;
* Participation in other interventional clinical studies within 30 days prior to Day 1;
* Other known co-existing malignancies except non-melanoma skin cancer and carcinoma in situ of the uterine cervix, unless definitively treated and proven no evidence of recurrence for 5 years;
* Any somatic or psychiatric disease/condition or abnormal laboratory test that in the opinion of the investigator, may interfere with the objectives and assessments of the study; or
* Unable to comply with the requirements of the study protocol or be unsuitable for the study for any reason, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of the objective response rate by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. | 24 months after last dose administration
  The morphological imaging (CT/MRI) will be done before therapy and selected time points before therapy cycle to determine changes in the size of target lesions.
Number of patients with treatment-related adverse events as assessed by CTCAE v.4.0 | 24 months after last dose administration
  To assess the safety and tolerability of 212Pb-DOTAMTATE

SECONDARY OUTCOMES:
Measurement of the Median Progression free survival (mPFS) | 24 months after last dose administration
  PFS will be defined as the number of days from the first dose of 212Pb-DOTAMTATE to documented tumor progression per RECIST 1.1 criteria or death due to any cause.
Measurement of Overall Survival (OS) | 24 months after last dose administration
  OS will be defined as the number of days from the first dose of 212Pb-DOTAMTATE to the date of death due to any cause or the date of last contact (censored observations) at the data cut-off date.
Measurement of Time to Tumor Progression (TTP) | 24 months after last dose administration
  This measurement will determine the time from start of treatment with 212Pb- DOTAMTATE until disease progression.
To evaluate health-related quality of life (HRQL) using ECOG performance status | 24 months after last dose administration
  Changes in quality of life will be assessed relative to baseline.
  Eastern Cooperative Oncology Group (ECOG) is designed to measure how cancer affects subject's daily life and is assessed using 0-5 scale.
To evaluate health-related quality of life (HRQL) using HRQL questionnaire EORTC QLQ-C30 | 24 months after last dose administration
  Changes in quality of life will be assessed relative to baseline.
  European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 is a self-assessed questionnaire that consists of 30 questions designed to measure varying types of functioning, symptoms and overall health/quality of life. It is assessed using either a 4-point scale or 7-point scale, depending on the question.
To evaluate health-related quality of life (HRQL) using HRQL questionnaire EORTC QLQ-G.I.NET21 | 24 months after last dose administration
  Changes in quality of life will be assessed relative to baseline.
  European Organisation for Research and Treatment of Cancer (EORTC) QLQ-G.I.NET21 is a self-assessed questionnaire that consists of 51 questions designed to assess symptoms or problems. It is assessed using a 4-point scale.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Louisiana State University (LSU) Health Sciences Center - New Orleans, Metairie, Louisiana
  - Excel Diagnostics and Nuclear Oncology Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No